CLINICAL TRIAL: NCT05924594
Title: A Phase 3, Dose-Optimized, Double-Blind, Randomized, Placebo-Controlled, Parallel Efficacy and Safety Laboratory Classroom Study in Children (6-12) With Attention-Deficit/Hyperactivity Disorder (ADHD) Using CTx-1301 (Dexmethylphenidate)
Brief Title: Phase 3 Efficacy and Safety Laboratory Classroom Study in Pediatrics (6-12) With ADHD Using CTx-1301
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Continuation of the study is not required for NDA submission via the 505(b)(2) pathway
Sponsor: Cingulate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTx-1301-004
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: ADHD; ADHD - Combined Type; Attention Deficit Hyper Activity; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder With Hyperactivity; Attention Deficit Hyperactivity Disorder Combined; Attention-deficit Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Experimental: 6.25mg CTx-1301 (Dexmethylphenidate tablet) (Experimental): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg. The starting dose for all subjects at Day 0 is 6.25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 6.25mg
- Experimental: 12.5mg CTx-1301 (Dexmethylphenidate tablet) (Experimental): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg. The starting dose for all subjects at Day 0 is 6.25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 6.25mg; Drug: CTx-1301 - Dexmethylphenidate 12.5mg
- Experimental: 18.75mg CTx-1301 (Dexmethylphenidate tablet) (Experimental): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg. The starting dose for all subjects at Day 0 is 6.25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 6.25mg; Drug: CTx-1301 - Dexmethylphenidate 12.5mg; Drug: CTx-1301 - Dexmethylphenidate 18.75mg
- Experimental: 25.0mg CTx-1301 (Dexmethylphenidate tablet) (Experimental): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg. The starting dose for all subjects at Day 0 is 6.25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 6.25mg; Drug: CTx-1301 - Dexmethylphenidate 12.5mg; Drug: CTx-1301 - Dexmethylphenidate 18.75mg; Drug: CTx-1301 - Dexmethylphenidate 25.0mg
- Experimental: 31.25mg CTx-1301 (Dexmethylphenidate tablet) (Experimental): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg. The starting dose for all subjects at Day 0 is 6.25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 6.25mg; Drug: CTx-1301 - Dexmethylphenidate 12.5mg; Drug: CTx-1301 - Dexmethylphenidate 18.75mg; Drug: CTx-1301 - Dexmethylphenidate 25.0mg; Drug: CTx-1301 - Dexmethylphenidate 31.25mg
- Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet) (Experimental): All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg. The starting dose for all subjects at Day 0 is 6.25mg. Each subject is expected to be on their optimal dose for 2 sequential weeks prior to the randomization phase. Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: CTx-1301 - Dexmethylphenidate 6.25mg; Drug: CTx-1301 - Dexmethylphenidate 12.5mg; Drug: CTx-1301 - Dexmethylphenidate 18.75mg; Drug: CTx-1301 - Dexmethylphenidate 25.0mg; Drug: CTx-1301 - Dexmethylphenidate 31.25mg; Drug: CTx-1301 - Dexmethylphenidate 37.5mg
- Placebo Comparator: Placebo (Placebo Comparator): Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomization phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTx-1301 - Dexmethylphenidate 6.25mg — All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg of CTx-1301.
  Other Names: 6.25mg CTx-1301 (Dexmethylphenidate tablet)
  Arms: Experimental: 12.5mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 18.75mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 25.0mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 31.25mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 6.25mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 12.5mg — All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg of CTx-1301.
  Other Names: 12.5mg CTx-1301 (Dexmethylphenidate tablet)
  Arms: Experimental: 12.5mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 18.75mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 25.0mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 31.25mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 18.75mg — All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg of CTx-1301.
  Other Names: 18.75mg CTx-1301 (Dexmethylphenidate tablet)
  Arms: Experimental: 18.75mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 25.0mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 31.25mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 25.0mg — All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg of CTx-1301.
  Other Names: 25.0mg CTx-1301 (Dexmethylphenidate tablet)
  Arms: Experimental: 25.0mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 31.25mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 31.25mg — All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg of CTx-1301.
  Other Names: 31.25mg CTx-1301 (Dexmethylphenidate tablet)
  Arms: Experimental: 31.25mg CTx-1301 (Dexmethylphenidate tablet); Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
Drug: CTx-1301 - Dexmethylphenidate 37.5mg — All subjects will be titrated to their optimal dose during the dose-optimization phase. Possible doses are 6.25mg, 12.5mg, 18.75mg, 25.0mg, 31.25mg, or 37.5mg of CTx-1301.
  Other Names: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
  Arms: Experimental: 37.5mg CTx-1301 (Dexmethylphenidate tablet)
Drug: Placebo — Subjects will be randomized (1:1) to their optimal dose or placebo in the 7-day, double-blind, randomized phase.
  Arms: Placebo Comparator: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of CTx-1301 in children (6-12) with ADHD in a laboratory classroom setting.

DETAILED DESCRIPTION:
A Phase 3, dose-optimized, randomized, double-blind, placebo-controlled, dose-optimized, parallel efficacy and safety laboratory classroom study in children (6-12) with ADHD.

The study will be comprised of a screening period, a dose-optimization phase, a double-blind randomized phase, and a safety follow-up phase. Subjects will undergo a screening visit prior to entering into a 8-week dose-optimization phase. During the dose-optimization phase, subjects will have weekly visits and will be titrated to doses ranging between 6.25mg-37.5mg of CTx-1301. Eligible subjects will be randomized phase to their optimal dose or placebo in a 1:1 ratio at the end of Visit 10 completing the practice laboratory classroom study. Subjects will take their assigned/randomized dose over the following 7-day period. On the 7th days subjects will complete the full laboratory classroom study. The duration of the full laboratory classroom study will be approximately 15 hours. Subjects will have an in-clinic safety follow-up visit within 7 days after the full classroom day.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 6 and 12 years of age (inclusive) at the time of consent.
2. Subject must have a body weight between the 5th and 95th percentile (≥5th percentile and ≤95th percentile) for their respective age and sex.
3. Subject is unsatisfied with his/her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects who are naïve to pharmacological therapy for ADHD or are newly diagnosed with ADHD is permitted.
4. Females of childbearing potential must have a negative serum b-human chorionic gonadotropin pregnancy test at Screening. Child-bearing potential is defined as any female who has had their first period or is 12 years or older (or will be 12 during the study). Female of childbearing potential or that become child-bearing potential during the study must agree to use a highly effective, medically acceptable form of birth control for 30 days prior to Screening until at least 30 days after the last dose of study drug. Alternatively, subject may remain abstinent until at least 30 days after the last dose of study drug. Episodic abstinence is not reliable to avoid pregnancy, so is not considered a highly effective contraceptive method. Investigator discretion should use judgement and familiarity with the subject's "preferred and usual lifestyle" to assess if reporting of abstinence may be trusted to achieve required effectiveness. Male subjects with female partners must agree at Screening to remain abstinent or agree to use an effective and medically acceptable form of birth control from Screening to 90 days after the last dose of study drug.
5. Subject must be in general good health defined as absence of any clinically significant abnormalities as determined by the Investigator based on physical and neurological examinations, vital signs, ECGs, medical history, and safety laboratory tests at screening. If any of the exams or tests are not within the laboratory reference range, the Investigator must assess and determine if clinically significant.
6. Subject's intellectual function is at an age-appropriate level, as deemed by the Investigator.
7. Subjects need to be able to perform at least the basic level of problems on the PERMP pre-test with at least 5.5 questions answered correctly per minute performed at Visit 2.
8. Subject must meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for the primary diagnosis of ADHD or any of the three presentations (combined, inattentive, or hyperactive/impulsive presentation) upon clinical evaluation and confirmed by the MINI International Neuropsychiatric Interview of Children and Adolescents (MINI-KID). The MINI-KID should also be used to evaluate any other psychotic disorders.
9. Subject must score 28 or higher on the ADHD-RS-5 scale at the screening visit (Visit 1) and Baseline visit (Visit 2). For subjects requiring washout of ADHD medications, adequate washout of stimulant ADHD medications will be defined as no medication for the previous 5 days. Adequate washout of non-stimulant ADHD medications will be defined as no medication for the previous 21 days.
10. Subject must have a score of 4 (moderately ill) or higher on the clinician-administrated Clinical Global Impressions-Severity (CGI-S) scale at screening (Visit 1). For subjects requiring washout of ADHD medications, adequate washout of stimulant ADHD medications will be defined as no medication for the previous 5 days. Adequate washout of non-stimulant ADHD medications will be defined as no medication for the previous 21 days.
11. Subject must be able and willing to wash out of stimulant ADHD medications (except study drug as indicated per protocol), including herbal medication, from 5 days prior to the start of the dose optimization phase (Visit 2) and for the duration of the entire study, defined as completion of the safety follow-up visit. Additionally, subject must be able and willing to wash out from non-stimulant ADHD medications 21 days prior to the start of the dose optimization phase (Visit 2) and for the duration of the entire study, defined as completion of the safety follow-up visit.
12. Subject and parents/legal guardians, and/or caregiver (if applicable) must be able to read, write, speak, and understand English and be able to communicate with the Investigator and study coordinator in a satisfactory fashion and complete any study-related materials. Subject and parents/legal guardians, and/or caregivers (if applicable) must plan to be available for the entire duration of the study.
13. One or more of the parents/legal guardians, or caregivers of the subject must voluntarily give written permission for him/her to participate in the study.
14. Subject must provide written assent prior to study participation
15. Subject, subject's parents/legal guardians, and/or caregivers (if applicable) must understand and be willing and able to comply with study procedures as well as the visit schedule. If the subject is cared for by a caregiver for relevant portions of the day, the caregiver may be more suitable for certain assessments, and the caregiver will need to agree to the applicable procedures and visits. The most appropriate assessor should be determined prior to the double-blind, randomized, efficacy portion. The assessor for each individual subject should be the same assessor throughout the double-blind, randomized, efficacy portion of the study.
16. Subject must be able to swallow the CTx-1301 tablet as evidenced by ability to swallow a similar size tablet (placebo) at screening.

Exclusion Criteria:

1. If female and of child-bearing potential, the subject must not be pregnant or breastfeeding at any time during the study or for 30 days following the completion of the study. If of child-bearing potential, urine hCG tests will be administered at protocol-specified time points. Any positive pregnancy test during the study will exclude them from further participation in the study.
2. Subject has any psychiatric diagnosis of bipolar I or II disorder, major depressive disorder, conduct disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, obsessive-compulsive disorder, eating disorder, anxiety disorder (including generalized anxiety disorder), any history of psychosis, autism spectrum disorder, a history of motor or vocal tics or Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances, or any other diagnosis/significant medical history that at the discretion of the Investigator excludes the subject from entry into the study.
3. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder (excluding febrile seizures), vascular disorder, potential CNS-related disorders that might occur in childhood, or history of persistent neurological symptoms related to a serious head injury.
4. Subject has any clinically significant and/or unstable/uncontrolled medical abnormality, chronic medical condition, persistent neurological symptoms, history of cardiovascular abnormality, abnormalities of respiratory, hepatic, gastrointestinal, renal, or any disorder or history of a condition that would impact or interfere with drug absorption, distribution, metabolism, or excretion during the study or may interfere with the subject's ability to participate in the study.
5. Subject has family history of early cardiovascular disease or sudden death.
6. Subject has any history of attempted suicide, clinically significant suicidal ideation based on the Columbia Suicide Severity Rating Scale (C-SSRS) assessment, or answers "yes" to "Suicidal Ideation" item 4 or 5 of any lifetime history on the C-SSRS Children's Lifetime/Recent assessment at screening.
7. Subject has a known primary sleep disorder (e.g., sleep apnea, narcolepsy, etc.)
8. If the subject's blood pressure is < 90th percentile for their age, sex, and height, the single read is sufficient. If the subject's blood pressure is ≥ 90th percentile, two additional reads will be taken, and the three reads will be averaged. If the average of the three readings is ≥ 95th percentile at screening they will be excluded.
9. Subject is considered treatment refractory by the Investigator or is intolerant to stimulant ADHD medication.
10. Any use of anticonvulsants currently or within the past 2 years.
11. Uncontrolled thyroid disorder indicated by thyroid stimulating hormone (TSH) ≤0.8 x the lower limit of normal (LLN) or ≥ 1.25 x the upper limit of normal (ULN) from the reference laboratory.
12. Subject has first-degree relatives (biological parent or sibling) with a history of schizophrenia, schizoaffective disorder, bipolar I disorder, or bipolar II disorder.
13. Subject has history of substance abuse or shows evidence of substance or has a positive urine drug screen at screening and/or baseline. Subjects with positive drug screens may be allowed to continue in the study if the result of the positive drug screen is from prescribed medications and the subject is willing to washout of the medication as required per protocol.
14. Previous treatment experience/exposure to CTx-1301.
15. Subject has a history of allergic reaction or sensitivity to methylphenidate, dexmethylphenidate, or any other substance contained in CTx-1301 or the placebo drug.
16. Subject has participated in a classroom study within 6 months prior to the start of Screening or has participated in any other clinical study with an investigational drug/product within 30 days prior to Screening or is currently participating in another clinical study.
17. Subject's family anticipates a move outside the geographic range of the investigative site during the duration of the study period or plans on travel that would not allow compliance to the protocol during the study period.
18. Subject is unsuitable in any other way, to participate in the study, as determined by the Investigator.
19. Subject is a family member of an employee at the study center, of the investigator, or those with direct involvement in the proposed study under the direction of that investigator or study center.
20. Subjects that are siblings are not allowed to be in the same cohort.

Eligibility Criteria (end of dose-optimization phase)

Subjects will be required to meet the following additional eligibility criteria at the end of the dose-optimization phase (Visit 10) to enter into the double-blind, randomized phase. These criteria are based on the efficacy and safety observed over the 8-week dose-optimization period.

1. A minimum of 2 weeks on optimal dose
2. A reduction of greater than or equal to 30% reduction of the ADHD-RS-5 from Visit 2 to Visit 10 (plus or minus 3 days) during the dose-optimization phase.
3. A CGI-I score of 1 or 2 points ("Very much improved" or "Much improved") at the end of the dose optimization phase (Visit 10 (plus or minus 3 days)).
4. Acceptable tolerability of the optimized CTx-1301 dose during the optimization phase (Visit 2 - Visit 10 (plus or minus 3 days)).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (pre-dose measured at Day 63) of the Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale (SKAMP)-combined scores collected across the 14-hour classroom day. | Baseline (pre-dose at Day 63) and at 0.5, 1, 3, 6, 9, 12, 13 and 14 hours post-dose during the full classroom day on Day 63.
  The Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) is a validated rating of subjective impairment of classroom behaviors. It is a 13-item scale, grouped by subcategories of attention, deportment, quality of work, and compliance. Subjects are rated according to a 7-point scale of impairment, with 0 being none and 6 being maximal impairment. A higher SKAMP score signifies greater impairment.

SECONDARY OUTCOMES:
Secondary Outcome Measure - Laboratory Classroom Onset and Duration | Baseline (pre-dose at Day 63) and at 0.5, 1, 3, 6, 9, 12, 13 and 14 hours post-dose during the full classroom day on Day 63.
  Onset and duration of the clinical effect of CTx-1301 during the 14-hour classroom day.
  The Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) is a validated rating of subjective impairment of classroom behaviors. It is a 13-item scale, grouped by subcategories of attention, deportment, quality of work, and compliance. Subjects are rated according to a 7-point scale of impairment, with 0 being none and 6 being maximal impairment. A higher SKAMP score signifies greater impairment.
Secondary Outcome Measure - CGI-S | Baseline (pre-dose measured at Day 0) to Day 63 (approximately 9 weeks).
  Change from baseline (pre-dose measured at Day 0) of Clinical Global Impression - Severity (CGI-S) scores to CGI-S at Day 63.
  The CGI-S is a clinician-rated scale that evaluates the severity of ADHD symptoms on a scale from 1 (not at all ill) to 7 (among the most severely ill).
Secondary Outcome Measure - SKAMP | Baseline (pre-dose at Day 63) and at 0.5, 1, 3, 6, 9, 12, 13 and 14 hours post-dose during the full classroom day on Day 63.
  Mean of the changes from baseline (pre-dose measured at Day 63) of the Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale (SKAMP)-Deportment scores (SKAMP-D) and (SKAMP)-Attention scores (SKAMP-A) collected across the 14-hour classroom day.
  The Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) is a validated rating of subjective impairment of classroom behaviors. It is a 13-item scale, grouped by subcategories of attention, deportment, quality of work, and compliance. Subjects are rated according to a 7-point scale of impairment, with 0 being none and 6 being maximal impairment. A higher SKAMP score signifies greater impairment.
Secondary Outcome Measure - PERMP-C | Baseline (pre-dose at Day 63) and at 0.5, 1, 3, 6, 9, 12, 13 and 14 hours post-dose during the full classroom day on Day 63.
  Change from baseline (pre-dose measured at Day 63) of the Permanent Product Measure of Performance - Correct (PERMP-C) scores collected across the 14-hour classroom day.
Secondary Outcome Measure - CGI-I | Baseline (pre-dose at Day 63) compared to Day 63
  While CGI-I will be analyzed using the mean change from Baseline (pre-dose at Day 63) compared to Day 63

OTHER OUTCOMES:
Exploratory Endpoints | • Evaluate overall treatment experience of subjects who have ever taken an ADHD stimulant medication prior to screening (Visit 1) using the entrance questionnaire. • Evaluate overall treatment experience of CTx-1301 at Day 56 (end of dose optimization)
  Exploratory efficacy endpoints will evaluate the quality and satisfaction of prior medications and of CTx-1301 during screening and D56

CONTACTS AND LOCATIONS:
Overall Officials: Matt Brams, MD, Study Director — Cingulate
Locations (3):
- United States (3):
  - Accel Research Sites, Maitland, Florida
  - Center for Psychiatry & Behavioral Medicine, Las Vegas, Nevada
  - Coastal Carolina Research Center, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
Overall study data as required by FDAAA801 will be shared upon completion of the study